CLINICAL TRIAL: NCT06368934
Title: Sub-lobectomy for IDH Wild-type and TERT Promoter Mutant Glioblastoma: A Prospective, Interventional, Multicenter, Randomized Controlled Trial
Brief Title: Sub-lobectomy for IDH Wild-type and TERT Promoter Mutant Glioblastoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jinsong Wu, Chief Physician, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2024-011
Record Dates: First submitted 2024-02-27; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Glioma; Glioblastoma
MeSH Terms: conditions — Glioma; Glioblastoma

STUDY DESIGN:
Intervention Model Description: Type of study: randomized parallel controlled, open-label, multicenter clinical trial.
  Interventions: the intervention group was to receive frontal, temporal, parietal, and occipital sub-lobotomies that met anatomical criteria, and the control group was to receive imaging total resection (T1-enhanced borders) that met the Response Assessment in Neuro-Oncology (RANO) criteria.
  Randomization The control group and intervention group were equal in size. Following intraoperative pathological diagnosis, participants were randomly assigned using a centralized randomization system known as the Interactive Web Response System (IWRS). Stratification factors included preoperative age brackets of [18-65] and (65-80), gender (male or female), and tumor site in the frontal, temporal, parietal, and occipital lobes.
Who Masked: Participant
Masking Description: This study employed a single-blind approach whereby the participants were unaware of the kind of surgical resection they were receiving.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group was to receive frontal, temporal, parietal, and occipital sub-lobotomies that met anatomical criteria.
  Interventions: Procedure: sub-lobectomy
- The control group (Other): The control group was to receive imaging total resection (T1-enhanced borders) that met RANO criteria.
  Interventions: Procedure: imaging total resection

INTERVENTIONS:
Procedure: sub-lobectomy — Combined with previous research and our team's precise neurosurgery concept, we define the surgical strategy based on lobectomy and further preserving the brain parenchyma in functional areas according to anatomical landmarks and electrophysiological boundaries as sub-lobectomy.
  Arms: The intervention group
Procedure: imaging total resection — Imaging total resection (T1-enhanced borders) will met the RANO criteria
  Arms: The control group

SUMMARY:
Glioblastoma is recognized as the most common and aggressive form of primary malignant brain tumor, with treatment options that are limited and prognosis that is extremely poor, showing median progression-free survival of 12 months and median overall survival of less than 18 months. Surgical resection plays a critical role in the treatment, with the extent of resection significantly impacting patient outcomes. Historical approaches to surgical resection have evolved, moving from radical strategies to more conservative ones that aim to preserve normal brain function while removing the tumor as completely as possible. Recent studies have suggested that increasing the extent of surgical resection, particularly along the T2 FLAIR border rather than the traditional T1-enhanced border, can significantly improve patient prognosis. There is, however, a lack of consensus on the optimal surgical approach, and the heterogeneity of tumors presents challenges in standardizing surgical strategies. Extended resection has been shown to prolong survival, and novel intraoperative molecular diagnostics have emerged to improve accuracy in tumor classification and prognosis. Building on these advancements, a multicenter, prospective, randomized controlled trial is proposed to evaluate the efficacy of sub-lobectomy in treating IDH wild-type/TERTp-mutant glioblastoma, aiming to improve evidence levels and establish standardized surgical practices for this devastating disease.

DETAILED DESCRIPTION:
Glioblastoma is the most prevalent and aggressive type of primary malignant brain tumor[1]. Treatment options are limited and often include surgical resection followed by radiation therapy or electric field therapy[2]. Prognosis is very poor, with median progression-free survival of only 12 months and median overall survival of less than 18 months. The 5-year survival rate is a mere 12% [3].

Surgical resection is fundamental to treating patients with glioblastoma, and the extent of resection directly impacts patient prognosis [4]. Professor William Stewart Halsted, a renowned surgeon, historically championed "radical" surgical resection as a means of controlling tumours [5]. Nevertheless, the majority of neurosurgeons disagreed with this view because of the disruption to normal brain function caused by extreme surgery. However, in 1928, Professor Walter Dandy reported five patients with gliomas who underwent right hemispherectomy [6]. These patients showed no significant neurological impairment except for left hemiparesis. Even though no grave complications arise from the complete resection of the nondominant hemisphere, it did not seem to enhance the patients' prognosis either. Only one out of these five patients survived for 3.5 years, and eventually, all of them passed away due to gliomas. After this, the radical surgical strategy of enlarging the resection margin around gliomas was challenged, and neurosurgeons aimed to achieve total resection of imaging gliomas, based on the principle of removing tumour tissue with an abnormal signal on MRI while preserving normal brain function.

Notably, with respect to the complete surgical removal of glioblastoma, the T1-enhanced borders of MRI imaging were commonly used as a criterion in the past. However, various retrospective studies reveal that increasing the extent of surgical resection significantly improves patient prognosis (median survival from 9.8 to 15.2 months) [7]. However, a recent study conducted retrospectively discovered that resection along the T2 FLAIR border advanced the prognosis of patients with glioblastoma even further compared to resection along the T1 enhancing border (median survival from 11.6 to 31.7 months) [8]. Another study discovered that performing a sub-lobectomy on glioblastoma patients could enhance their prognosis (median survival from 18.7 to 44.1 months) in comparison to T2 FLAIR border resection, as long as normal brain function is not affected [9]. Nonetheless, there remains a lack of consensus in the academic community regarding the optimal surgical resection strategy for glioblastoma patients (such as T1 enhancing border, T2 FLAIR border, sub-lobectomy). In addition, the significant heterogeneity in tumour location, size, infiltration extent, and anatomical proximity across different patients makes it difficult to standardise imaging border resection as an "individualised" surgical approach. This places greater demands on the surgical capabilities and knowledge of clinicians in clinical settings. Furthermore, it also introduces multiple confounding factors that hinder the advancement of interventional clinical research.

Therefore, we have thoroughly reviewed recent studies to investigate the prognosis of glioblastoma patients following extended resection. The majority of studies analyzed the prognostic benefits of extended resection beyond T1 enhancement compared to gross total tumor resection, while a few studies evaluated the difference between sub-lobectomy and gross total tumor resection. Extended resection beyond the T1 enhancement region was discovered to prolong the survival of glioblastoma patients, with the prognostic benefits of sub-lobectomy proving significantly pronounced and not associated with further neurological impairment [9]. Previous studies have several limitations. Firstly, they are predominantly retrospective, leading to issues with selection bias and retrospective memory bias, among other factors. Furthermore, many of these studies lack a balanced control group. Secondly, factors such as a small number of patient cases, short follow-up time, and poor quality control of follow-up have also contributed to their low level of evidence [10]. Furthermore, the classification for glioblastoma were updated in 2021. Patients with gliomas who were included in these studies also await further evaluation to clarify their diagnosis.

Previous studies on the correlation between surgical resection and prognosis of glioblastoma were retrospective due to the absence of molecular pathology. Intraoperative frozen pathology cannot provide real-time diagnosis of glioblastoma. Therefore, molecular testing is crucial for accurate staging and diagnosis. According to the 5th edition of World Health Organization Central Nervous System tumors classification, patients diagnosed with glioblastoma (IDH wild-type) had IDH wild-type adult diffuse glioma accompanied by tissue necrosis, vascular hyperplasia, TERT promoter mutation, +7/-10, or epidermal growth factor receptor (EGFR) amplification [17]. TERT promoter mutation, which is the most frequent hotspot mutation observed in glioblastomas, is present in almost 80% of patients with glioblastoma mutations [18]. We have conducted a range of innovative studies regarding intraoperative rapid integrated diagnosis of gliomas. Our works include ①simplified integrated diagnostic system for human gliomas that is based on a combination of IDH, TERT, and histopathology. ②We have also developed an accurate method for detecting IDH and TERT mutations through the use of locked nucleic acid-amplification refractory mutation system fluorescence polymerase chain reaction (PCR). ③We have optimized the DNA extraction process and reduced the detection cycle as well. ④Conducting multi-center, prospective clinical trials to verify the feasibility of intraoperative rapid molecular testing. In summary, through combining intraoperative frozen pathology, our technique allows for precise diagnosis of glioblastoma (IDH wild-type) with TERT promoter mutations within 35 minutes intraoperatively, with a sensitivity and specificity of 100.0% when compared with postoperative sequencing data. Furthermore, our prior retrospective study found that a higher degree of surgical resection greatly improved the prognosis of glioblastoma with IDH wild-type/TERTp-mutated, and that sub-lobectomy conferred a more significant prognostic benefit.

Therefore, building on previous work and knowledge in our field, we will conduct a multicenter, prospective, randomized controlled trial to evaluate the efficacy of sub-lobectomy in the treatment of IDH wild-type/TERTp-mutant glioblastoma. Our study aims to enhance the level of evidence, while also establishing a standardized surgical strategy for glioblastoma.

ELIGIBILITY:
Inclusion Criteria:

1. Eligible patients are aged between 18 and 80, have newly diagnosed high-grade diffuse adult-type gliomas, and have not received any other treatment besides puncture biopsy.
2. Preoperative KPS score ≥70.
3. Enhanced MRI can be tolerated.
4. Sign the informed consent form.
5. Patients with supratentorial gliomas and lesions confined to the unilateral frontal, temporal, parietal, and occipital lobes are included.
6. Imaging total resection can be completed after preoperative imaging evaluation.
7. The intraoperative integrative diagnosis was IDH wild-type high-grade glioma with TERT promoter mutation.

Exclusion Criteria:

1. The tumor involves the anterior central gyrus, posterior central gyrus, nigral gyrus, limbic lobe, corpus callosum, basal ganglia, and lateral ventricles.
2. The tumor involves 2 or more lobes of the brain;
3. Developing severe systemic diseases such as renal insufficiency, hepatic insufficiency, cardiac insufficiency, etc.
4. Previously, the patient had experienced other types of malignant tumours.
5. Developing other brain diseases, such as Parkinson's or Alzheimer's disease.
6. Simultaneously participating in other clinical trials.
7. Expected survival is less than 3 months.
8. Not receiving Stupp protocol after surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 326 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival | From date of randomization until the date of first documented progression, assessed up to 36 months
  Progression-free Survival (PFS) in patients with IDH wild-type/TERTp-mutant glioblastoma in the sub-lobectomy group and in the imaging total resection (T1-enhanced border) group.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization until the date of death from any cause, assessed up to 36 months
  Overall Survival (OS) in patients with IDH wild-type/TERTp-mutant glioblastoma in the sub-lobectomy group and in the imaging total resection (T1-enhanced border) group.

OTHER OUTCOMES:
Postoperative quality of life | up to 6 months
  Using Karnofsky Performance Scale (KPS) to evaluate for postoperative quality of life.
Adverse effects | up to 6 months
  The Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE™) scale was used to assess adverse effects.
Cognitive function | up to 3 months
  The cognitive function will be assessed by Mini-mental State Examination (MMSE) scale.
Language function | up to 3 months
  The language function will be assessed by aphasia examination of chinese.
Limb muscle strength | up to 3 months
  The limb muscle strength will be assessed by Manual Muscle Test (MMT).

CONTACTS AND LOCATIONS:
Locations (1):
- Hushan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] [1]. Weller M, Wick W, Aldape K, et al. Glioma. Nature Reviews Disease Primers 2015;1:15017. [2]. Schaff Lauren R,Mellinghoff Ingo K,Glioblastoma and Other Primary Brain Malignancies in Adults: A Review.[J] .JAMA, 2023, 329: 574-587. [3]. Xiong Z, Luo C, Wang P, Hameed NUF, Song S, Zhang X, Wu S, Wu J, Mao Y. The Intraoperative Utilization of Multimodalities Could Improve the Prognosis of Adult Glioblastoma: A Single-Center Observational Study. World Neurosurg. 2022 Sep;165:e532-e545. [4]. 罗宸, 吴帅, 吴劲松. 分子病理指导下的脑胶质瘤手术的研究进展.中华神经外科杂志, 2021, 37(9). 952-956. [5]. Halsted WS: I. The results of operations for the cure of cancer of the breast performed at the Johns Hopkins Hospital from June, 1889, to January, 1894. Ann Surg 20:497-555,1894. [6]. Dandy WE: Removal of right cerebral hemisphere for certain tumors with hemiplegia. J Am Med Assoc 90:823-825, 1928. [7]. Li YM, Suki D, Hess K, Sawaya R: The influence of maximum safe resection of glioblastoma on survival in 1229 patients: Can we do better than gross-total resection? J Neurosurg 124:977-988, 2016. [8]. Molinaro Annette M,Hervey-Jumper Shawn,Morshed Ramin A et al. Association of Maximal Extent of Resection of Contrast-Enhanced and Non-Contrast-Enhanced Tumor With Survival Within Molecular Subgroups of Patients With Newly Diagnosed Glioblastoma.[J] .JAMA Oncol, 2020, 6: 495-503. [9]. Roh Tae Hoon,Kang Seok-Gu,Moon Ju Hyung et al. Survival benefit of lobectomy over gross-total resection without lobectomy in cases of glioblastoma in the noneloquent area: a retrospective study.[J] .J Neurosurg, 2019, 132: 895-901. [10]de Leeuw CN, Vogelbaum MA. Supratotal resection in glioma: a systematic review. Neuro-Oncol. 2019;21(2):179-188. [11] Pessina F, Navarria P, Cozzi L, Ascolese AM, Simonelli M, Santoro A, Clerici E, Rossi M, Scorsetti M, Bello L. Maximize surgical resection beyond contrast-enhancing boundaries in newly diagnosed glioblastoma multiforme: is it useful and safe? A single institution retrospective experience. J Neurooncol. 2017 Oct;135(1):129-139. [12] Glenn CA, Baker CM, Conner AK, Burks JD, Bonney PA, Briggs RG, Smitherman AD, Battiste JD, Sughrue ME. An Examination of the Role of Supramaximal Resection of Temporal Lobe Glioblastoma Multiforme. World Neurosurg. 2018 Jun;114:e747-e755. [13] Salah M. Hamada, Ahmed H. Abou-Zeid. Anatomical resection in glioblastoma: extent of resection and its impact on duration of survival. 2016 The Egyptian Journal of Neurology, Psychiatry and Neurosurgery 1110-1083. [14] Di L, Shah AH, Mahavadi A, Eichberg DG, Reddy R, Sanjurjo AD, Morell AA, Lu VM, Ampie L, Luther EM, Komotar RJ, Ivan ME. Radical supramaximal resection for newly diagnosed left-sided eloquent glioblastoma: safety and improved survival over gross-total resection. J Neurosurg. 2022 May 27;138(1):62-69. [15] Schneider M, Potthoff AL, Keil VC, Güresir Á, Weller J, Borger V, Hamed M, Waha A, Vatter H, Güresir E, Herrlinger U, Schuss P. Surgery for temporal glioblastoma: lobectomy outranks oncosurgical-based gross-total resection. J Neurooncol. 2019 Oct;145(1):143-150. [16] Shah AH, Mahavadi A, Di L, Sanjurjo A, Eichberg DG, Borowy V, Figueroa J, Luther E, de la Fuente MI, Semonche A, Ivan ME, Komotar RJ. Survival benefit of lobectomy for glioblastoma: moving towards radical supramaximal resection. J Neurooncol. 2020 Jul;148(3):501-508. [17]. Louis DN, Perry A, Wesseling P, et al. The 2021 WHO Classification of Tumors of the Central Nervous System: a summary. Neuro-Oncology 2021;23:1231-51. [18]. Killela PJ, Reitman ZJ, Jiao Y, et al. TERT promoter mutations occur frequently in gliomas and a subset of tumors derived from cells with low rates of self-renewal. Proc Natl Acad Sci U S A 2013;110:6021-6. [19]. Ellingson BM, Wen PY, Cloughesy TF. Modified Criteria for Radiographic Response Assessment in Glioblastoma Clinical Trials. Neurotherapeutics. 2017 Apr;14(2):307-320.